CLINICAL TRIAL: NCT04438902
Title: A Prospective, Multi-center, Interventional Study of Osimertinib Combined With Anlotinib in Acquired EGFR T790M Mutated NSCLC Patients With Gradual Progression on Osimertinib Treatment
Brief Title: Osimertinib Combined With Anlotinib in EGFR T790M Mutated NSCLC Patients With Progression on Osimertinib Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Many patients can't tolerate the combination treatment due to adverse events.
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRAIN
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2021-06

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non-small-cell lung cancer; EGFR T790M; osimertinib; anlotinib; acquired resistance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open, single-arm, exploratory phase 2 trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osimertinib combined with anlotinib (Experimental)
  Interventions: Drug: osimertinib mesylate tablets and anlotinib hydrochloride capsules

INTERVENTIONS:
Drug: osimertinib mesylate tablets and anlotinib hydrochloride capsules — osimertinib mesylate tablets 80mg qd and anlotinib hydrochloride capsules 10mg qd day 1-14 of a 21-day cycle
  Other Names: TAGRISSO and FOCUS V

SUMMARY:
EGFR T790M gatekeeper mutation accounts for approximately 60% of acquired resistance to the first- or second-generation EGFR-TKI treatment. Osimertinib, a third-generation EGFR TKI, has become the standard therapy for NSCLC patients with acquired EGFR T790M mutation. However, acquired resistance to osimertinib is still inevitable and there is no established targetable agent currently. Thus, treatment strategy for patients with acquire resistance to osimertinib remains an urgent issue. In this study, we aimed to evaluate the efficacy of osimertinib combined with anlotinib in acquired EGFR T790M mutated NSCLC patients with gradual progression on osimertinib treatment.

DETAILED DESCRIPTION:
In current clinical practice, acquired resistance to osimertinib can be divided into three clinical modes: dramatic progression, gradual progression and local progression. For patients with gradual progression,there are various clinical explorations，including the continuation of osimertinib with chemotherapy or radiotherapy, osimertinib combined with antiangiogenic agents. In preclinical studies, an overactive vascular endothelial growth factor/vascular endothelial growth factor receptor (VEGF/VEGFR) pathway and tumour angiogenesis plays a crucial role in the resistance to EGFR-TKIs, and the dual targeting of both the VEGF and EGFR pathways may prevent resistance.

Anlotinib (AL3818) is an inhibitor targeting multiple receptor tyrosine kinases involved in tumour progression, especially VEGFR 2/3, PDGFRα/β and c-Kit. We suppose that the combination treatment of osimertinib and anlotinib may ameliorate acquired resistance to osimertinib.This is a multi-center, open, single-arm, exploratory phase 2 trial evaluating osimertinib combined with anlotinib in acquired EGFR T790M mutated NSCLC patients with gradual progression on osimertinib treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent, complete all study assessments and have complete medical record.
2. Age:18-75 years.
3. Histologically or cytologically confirmed diagnosis of local advanced or metastatic NSCLC.
4. Patients should be confirmed acquired EGFR T790M mutation and received osimertinib as the second line treatment, and they should have the following: (1) benefit from treatment with osimertinib initially ;(2) gradual progression on osimertinib treatment as defined by minor increment of tumor burden (≥10% but <20% in the sum of target lesions).
5. At least one measurable lesion as defined by lesions ≥10mm in long axis according to RECIST 1.1.

Exclusion Criteria:

1. Patients who will be or were involved in any other interventional antitumour clinical studies for locally advanced/metastatic NSCLC currently or previously.
2. Small cell lung cancer (including small lung cancer mixed with non-small cell lung cancer).
3. Patients at risk of bleeding.
4. Patients with renal dysfunction.
5. Uncontrolled severe hypertension.
6. Any concomitant condition evaluated by physicians which is not suitable for osimertinib or anlotinib treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | from the date of first dose of osimertinib until the date of disease progression，assessed up to 12 months.
  PFS is defined as the time from beginning of osimertinib to disease progression on combination treatment of osimertinib and anlotinib.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | from the date of combination of osimertinib and anlotinib, assessed up to 6 weeks.
  Objective Response Rate (ORR), is defined as the percentage of patients with complete response or partial response by investigator assessment as recorded in the CRF, which usually refer to Response Evaluation Criteria In Solid Tumours (RECIST) v1.1 in clinical practice.
Disease Control Rate (DCR) | from the date of combination of osimertinib and anlotinib, assessed up to 6 weeks.
  Disease Control Rate (DCR), is defined as the percentage of patients with complete response or partial response or stable disease by investigator assessment as recorded in the CRF, which usually refer to RECIST v1.1 in clinical practice.
Adverse events/Serious adverse events | From signing ICF to 30 days after the end of treatment.
  Incidence of Adverse Events (AEs): Incidence, severity and seriousness of adverse events, incidence of serious adverse events (SAEs), which usually be graded by CTCAE v5.0 based on current clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Yuehong Wang, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (2):
- China (2):
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Jiaxing College, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No
No plan to share participant data of the trial.